CLINICAL TRIAL: NCT05017181
Title: Assessment of Diagnostic and Prognostic VALue, Identification of bIological Correlates, and Determination of TEchnical Performance of Novel Metabolic and Microstructural MRI in PROstate Cancer
Brief Title: Novel MRI Assessment of Prostate Cancer VALIDATE-PRO
Acronym: VALIDATE-PRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 129237
Record Dates: First submitted 2021-05-17; First posted 2021-08-23 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
Keywords: MRI; biomarker; novel technique; cancer; validation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Prostatectomy digital histopathology metrics and biochemical stains for the prostatectomy arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BioVal: BioVal is a single site validation study to determine the histological correlates underpinning signals derived from 13C-pyruvate HYP-MRI in men with known prostate cancer scheduled for prostatectomy.
- ProVal: ProVal is a single site, prospective, longitudinal observational cohort study to determine the prognostic value of signals derived from VERDICT, Luminal Index MRI and 13C-pyruvate HYP-MRI in men with known early prostate cancer on active surveillance.
- TecVal: TecVal is a multi-site validation study to determine the inter-site repeatability and intra-site reproducibility of signals derived from VERDICT, Luminal Index MRI and 13C-pyruvate HYP-MRI in men with known prostate cancer.

SUMMARY:
For 50 years the diagnosis of prostate cancer has been with Prostate Specific Antigen (PSA) blood testing and prostate biopsy. However, this approach resulted in over-diagnosis, over-treatment and missed clinical important cancers. Multi-parametric MRI (mp-MRI) has provided a solution to some of these issues and the National Institute for health and Care Excellence has advocated the use of mp-MRI before biopsy in men with a suspicion for prostate cancer.

However, important challenges remain and the current way we pick up and assess prostate cancer can be improved. mp-MRI can miss significant cancer in around 11% of cases, 30% of positive MRI scans turn out not to have significant cancer at biopsy. Lastly, 34% of mp-MRI lesions are scored as in-determinant which sometimes makes decisions for further investigation and treatment unclear.

There are also difficulties predicting patients who will have progression of their disease or those who will not suffer harm from their cancer. Therefore the development of non-invasive tests and markers that can tell apart aggressive and non-aggressive disease would be extremely useful in deciding what treatment approach suits individual patients.

This study will investigate the use of three different novel MRI methods; Vascular, extracellular and restricted diffusion for cytometry in tumours (VERDICT), Luminal Imaging (LI) and hyperpolarised [1-13C]-pyruvate MRI (HYP-MRI). These scans help us to look at the microstructure as well as the metabolism of prostate tissue and may offer ways to better differentiate aggressive vs non-aggressive disease.

These scans will be performed in men with prostate cancer suitable for active surveillance at baseline and 1 year later to assess for prognostic indicators for progression in early prostate cancer.HYP-MRI will also be performed in men undergoing radical prostatectomy for validation of image findings and pathology. Whilst some men will have repeat scanning to asses for the repeatability of these techniques.

DETAILED DESCRIPTION:
PURPOSE AND DESIGN

The purpose of this study is to assess the ability of novel MRI techniques and their derived metrics in the diagnosis and prognostication of prostate cancer. Improving the diagnostic accuracy and investigating biomarkers with non- invasive MRI techniques have the promise of reducing unnecessary biopsies or radical treatment, as well as detecting those likely to progress at an earlier stage.

Vascular, Extracellular and Restricted Cytometry in Tumours (VERDICT) MRI

Diffusion-weighted imaging (DWI) is one of the most important sequences in mp-MRI of the prostate which reflects the diffusivity of water in cells and differs in cancerous tumour due to changes in cellular density, size, shape and arrangement. VERDICT is a novel framework which uses a more complex 3-compartment tissue model for diffusion of water; 1. Water trapped in cells, 2. Water in the vascular network and 3. Interstitial water. This allows us to make estimates of specific tissue properties such as the size and packing density of the cells, the vascular extracellular- extravascular space (EES) volume fractions. This methods is more biologically specific compared to conventional DWI. Studies in tumour xenograft models of colorectal cancer showed its ability to detect such known differences in the microstructure. At UCL we have applied VERDICT to the prostates of 78 men and were able to successfully differentiate between benign or clinically insignificant cancer and clinically significant tumours. This technique can be applied on commercially available MRI scanners and requires no additional contrast agents or requirements for the patient compared to conventional mp-MRI of the prostate.

Luminal Index (LI) MRI

Using a multi-echo T2 sequence we can differentiate between the relatively long T2 values of the luminal space and the short T2 values of the stromal and epithelial cells to estimate the fractional volume of water in each MR voxel, the luminal water fraction (LWF). Studies have shown a good correlation between LWF and histologically measure luminal fractional volume and hence promise to detect prostate cancer and predict Gleason score. Our refined local LI MRI sequence has been very good at differentiating clinically significant and non-significant tumours. This technique also requires no additional contrast agents or patient requirements to be completed.

Hyperpolarised [1-13C]-pyruvate MRI (HYP-MRI)

Cancer cell rely on enhanced glycolysis for their energy supply, a phenomenon known as the Warburg effect. This is a key discriminator of malignancy and normal tissues and has been successfully targeted with well-established imaging techniques such as Fluorodeoxyglucose (FDG) - Positron Emission Tomography (PET). HYP-MRI is able to image a part of this metabolic process in real-time. An injectable solution containing 13C labelled pyruvate which is hyperpolarised onsite in order to increase the eventual detectable signal. The naturally occurring metabolise pyruvate is converted to lactate with the attached 13C tag persisting enabling us to track the presence and conversion of pyruvate to lactate after the injection. It heralds the potential to differentiate tumours which are more likely to grow and metastasise from those which won't. This sequence requires an additional injection compared to standard mp-MRI and also uses an endorectal coil which is place inside the rectum for the duration of the scan.

The main objectives of this study are as follow and are addressed in three sub-studies:

* To biologically validate HYP-MRI with correlation against biological measurements in men undergoing radical prostatectomy (BioVal: 44 patients)
* Clinical validation of novel MRI techniques (VERDICT/LI/HYP-MRI) derived measurements for differentiating patients with aggressive (progressive) and indolent (non-progressive) prostate cancer in men entering active surveillance (ProVal: 120 patients)
* Technical validation of novel MRI techniques (VERDICT/LI/HYP-MRI) through assessment of repeatability metrics from derived parameters (TecVal: 20 patients)

ELIGIBILITY:
Inclusion Criteria:

* Men aged >18 years
* Pre-biopsy mp-MRI study performed within preceding 4 months
* Likert/PIRADS score 4-5/5 lesion and/or biopsy confirmed Prostate cancer
* Willing and able to provide written informed consent

Exclusion Criteria:

* Men who suffer with claustrophobia or are unable to have an MRI e.g. implantable defibrillator, brain aneurysm clips or other implant, severe obesity or unable to lay still for length of scan.
* Men with an impaired renal function (eGFR <30)
* Previous prostate radiotherapy/focal treatment
* Hormonal treatment for prostate cancer within preceding 3 months from consenting to the study.
* Dementia or other neurological condition meaning participant lacks the capacity to consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BioVal Cohort: Men scheduled for Prostatectomy
  ProVal Cohort: Men initiating active surveillance and treatment for low grade disease.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
ProVal Primary Objective | 3 years
  To determine the prognostic value of VERDICT metrics for risk classification of patients with early prostate cancer suitable for active surveillance.
  Quantitive value: fIC (intracellular (IC) volume fraction) among others within model.
ProVal Primary Objective | 3 years
  To determine the prognostic value of Luminal Index for risk classification of patients with early prostate cancer suitable for active surveillance.
  Quantitive value: Luminal index
ProVal Primary Objective | 3 years
  To determine the prognostic value of 13C-HYP-MRI for risk classification of patients with early prostate cancer suitable for active surveillance.
  Quantitive value: Lactate and pyruvate ratio parameters.
BioVal Primary Objective | 3 years
  To estimate the association of 13C-HYP-MRI derived quantitative metrics against histological features of prostate cancer.
  Quantitive value: Lactate and pyruvate ratio parameters.
BioVal Primary Objective | 3 years
  To estimate the association of 13C-HYP-MRI derived quantitative metrics against histological features of prostate cancer.
  Quantitive value: Gleason Grade
TecVal Primary Objective | 3 years
  Inter-site repeatability and intra-site reproducibility of signals derived from VERDICT, Luminal Index MRI and 13C-pyruvate HYP-MRI in men with known prostate cancer.
  Metric: Repeatability and reproducibility co-efficients

SECONDARY OUTCOMES:
ProVal Secondary Objective | 3 year
  To examine the effects of histological progression of prostate cancer on VERDICT and LI-MRI quantitative metrics To determine whether baseline imaging metrics can predict time to radiological progression.
  Metric: Gleason grade (used in combination with previous metrics discussed)

OTHER OUTCOMES:
ProVal Tertiary Objective | 3 years
  To link quantitative mpMRI, VERDICT MRI, LI-MRI and 13C-HYP-MRI quantitative features with molecular, genetic, epigenetic, transcriptomic and proteomic immune measurements made within patients recruited to the linked RECONCILE study.
  Metric: genetic, molecular and epigenetic measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Shonit Punwani, MD PhD, Principal Investigator — UCL
Locations (1):
- University College London, London, United Kingdom